CLINICAL TRIAL: NCT06705257
Title: EFFECT OF VARYING LEVELS OF PEEP ON PRETERM LUNG RECRUITMENT USING ELECTRICAL IMPEDANCE TOMOGRAPHY- FEASIBILITY STUDY
Brief Title: PEEP FOR LUNG RECRUITMENT IN PRETERM INFANTS-EIT STUDY
Acronym: [PEOPLE]
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Collaborators: The James Cook University Hospital Marton Road Middlesbrough TS4 3BW (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRAS [340081] - [PEOPLE]
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: PreTerm Neonate; Positive End Expiratory Pressure (PEEP); Lung Recruitment; Electrical Impedance Tomography (EIT)
Keywords: positive end expiratory pressure; PRETERM; Electrical Impedance Tomography
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Single arm. All the recruited preterm infants will undergo increasing and decreasing levels of PEEP and the effect of EIT with various PEEP levels will be studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single arm with increasing and decreasing PEEP levels (Experimental)
  Interventions: Diagnostic Test: Studying the effects of varying levels of PEEP using Electrical impedance tomography

INTERVENTIONS:
Diagnostic Test: Studying the effects of varying levels of PEEP using Electrical impedance tomography — Feasibility of using EIT, to study the effect of varying levels of PEEP/Continous distending pressure on lung recruitment as measured by changes in functional lung scores and silent spaces in preterm infants (<32 weeks) who are on mechanical ventilation or receiving primary or post extubation CPAP support.

SUMMARY:
Babies born early (under 32 weeks) are at risk of developing lung problems after birth. A major reason for this is that the lungs are not fully developed. Lungs of preterm babies will often collapse in between breathing due to lung immaturity. Applying gentle pressure, using nasal device through their nostril or through the breathing tube helps to prevent this lung collapse. This would help in air-oxygen going to lungs and also makes the babies breathing more comfortable. This gentle pressure is medically called as PEEP/CPAP and could be delivered by breathing machine (ventilator) and CPAP machine, collectively called as "continuous distending pressure (CDP)".

Those babies breathing on their own and receiving inadequate CDP would need more breathing support by placing them on breathing machine (ventilator). The longer the baby receives breathing machine support, higher chance of lung injury . Preterm infants who are already on breathing machine, providing sub optimal PEEP/CPAP could also lead to lung damage. Providing optimal PEEP/CPAP could prevent these negative outcomes. Currently there is not enough evidence to suggest optimal PEEP/CPAP in preterm infants. Neonatal units all around the world uses PEEP/CPAP ranging from 4 to 10cm H20 based on their unit practice. Currently available investigations provide limited one time information (e.g. Chest X-ray) regarding whether baby is receiving optimal PEEP/CPAP. Electrical Impedance Tomography (EIT) is a new technology which could provide better information regarding the pressure delivered. Also, this device would provide continuous information as if the clinicians are doing continuous chest X-ray but without any radiation. In this study, the team will assess the effect of different levels of PEEP/CPAP (4 to 10cm H20) on prevention of lung collapse using EIT. This would be studied in premature infants who are on breathing machine support and CPAP machine support.

ELIGIBILITY:
Inclusion criteria

1. Gestational age <32 weeks based on mother's last menstrual period or first trimester ultrasound dating.
2. Receiving either CPAP or mechanical ventilation respiratory support.
3. Informed written consent from one of the parents.
4. Within the first two weeks of life. Investigators pragmatically chose this period, as there could be considerable lung injury after the first two weeks of life, making it difficult to test our hypothesis. Also, this time period would allow parents to settle down with their stressful preterm delivery and investigators could approach anytime within the first two weeks of life.

Exclusion criteria

1. Major congenital malformations including congenital lung disease and congenital heart disease as ascertained by the medical team.
2. Infants diagnosed with pneumothorax i.
3. Receiving high frequency mechanical ventilation.
4. Infants with concerns of skin integrity.

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in EIT parameters | total study of 280 minutes
  Changes in End expiratory Lung Impedance scores
Changes in EIT parameters | 280minutes
  Changes in functional lung scores in percentage varying levels of CDP.
Changes in EIT | 280 minutes
  Changes in silence spaces with varying levels of CDP.

SECONDARY OUTCOMES:
Secondary outcomes | Total 280 minutes of study time
  Changes in oxygen saturation (SpO2 in percentage) during the study period.
Secondary outcome measure | Total study time of 280 minutes
  Changes in carbon dioxide levels as measured by transcutaneous carbon dioxide levels (TCO2) in kilopascal.
Secondary outcome | Total study time of 280 minutes
  Changes in fraction of inspiratory oxygen (Fio2) levels during the study.
Secondary outcome | Total study time of 280minutes
  Changes in blood pressure (if measured) during the study procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Mitchell, Study Director — South Tees NHS foundation trust

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the main study publication
Access Criteria: With valid study protocol and ethical approval.